CLINICAL TRIAL: NCT06948006
Title: An Open-label, Randomised, 2-arm, 3-period, 6-treatment Single-dose, Crossover Study Comparing the Pharmacokinetics of 2 Different Formulations of AZD4144, and Effect of Food and Omeprazole on the Pharmacokinetics of AZD4144 in Healthy Participants
Brief Title: A Study to Investigate the Relative Bioavailability of 2 Different Formulations of AZD4144, the Effect of Food and Omeprazole on the Pharmacokinetics of AZD4144 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D9441C00003
Record Dates: First submitted 2025-04-22; First posted 2025-04-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants
Keywords: Cardiorenal disease; Food effect; Proton-pump inhibitor; Pharmacokinetics; Tablet formulation
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: AZD4144 (Experimental): Participants will receive single doses of AZD4144 dose 1 as tablet formulation (Treatments A and B) and as an oral solution formulation (Treatment C) under fasted (Treatments A and C) and fed (Treatment B) conditions.
  Interventions: Drug: AZD4144
- Arm 2: AZD4144 + Omeprazole (Experimental): Participants will receive single doses of AZD4144 dose 2 tablet formulation under fasted (Treatment D) and fed (Treatment E) conditions and co-administered with omeprazole (Treatment F).
  Interventions: Drug: AZD4144; Drug: Omeprazole

INTERVENTIONS:
Drug: AZD4144 — Participants will receive AZD4144 orally.
Drug: Omeprazole — Participants will receive omeprazole orally.
  Arms: Arm 2: AZD4144 + Omeprazole

SUMMARY:
The main aim of this study to compare the pharmacokinetics (PK) of two formulations of AZD4144 and assess the effect of food and omeprazole on PK of AZD4144 in healthy participants.

DETAILED DESCRIPTION:
This is an open-label, randomized, single-dose, crossover Phase I study.

The study will comprise:

1. A Screening Period of 28 days.
2. Three Residential Periods
3. A final Follow-up period within 7 to 10 days after the last dose of study drug. There will be a minimum washout period of 7 days between each AZD4144 dose.

This study includes the following 2 arms:

Arm 1 consists of 3 treatments:

1. Treatment A: AZD4144 dose 1 as tablet (under fasted condition)
2. Treatment B: AZD4144 dose 1 as tablet (under fed condition)
3. Treatment C: AZD4144 dose 1 as an oral solution (under fasted condition)

Arm 2 consists of 3 treatments:

1. Treatment D: AZD4144 dose 2 as tablet (under fasted condition)
2. Treatment E: AZD4144 dose 2 as tablet (under fed condition)
3. Treatment F: Omeprazole once daily for 4 days, followed by a single dose of omeprazole along with a single dose of AZD4144 dose 2 as tablet (under fasted condition).

The participants will be randomised to one of the following treatment sequences:

Arm 1: ABC, BCA or CAB Arm 2: DEF or EDF

ELIGIBILITY:
Inclusion Criteria:

1. Signed the informed consent form before any study-related procedure.
2. Healthy male and female participants with suitable veins for cannulation or repeated venipuncture.
3. Negative pregnancy test for females at screening, first admission, and follow-up.
4. Females of childbearing potential must use highly effective contraception from first dose until 3 months after last dose.
5. Non-childbearing potential females must meet postmenopausal or surgical sterilization criteria.
6. Sexually active fertile males must use contraception from first dose until 3 months after last dose.
7. Body Mass Index (BMI) between 18-32 kg/m2 and weight ≥45 kg at screening and first admission.

Exclusion Criteria:

1. History of any clinically important disease or disorder that may put the participant at risk or influence study results.
2. History or presence of gastrointestinal, hepatic, or renal disease or any condition affecting drug absorption, distribution, metabolism, or excretion.
3. Any clinically important illness, medical/surgical procedure, or trauma within 4 weeks of randomization.
4. Active systemic bacterial, viral, or fungal infection within 14 days prior to dosing or presence of fever within 14 days prior to dosing.
5. Clinically significant serious active and chronic infections within 60 days prior to randomization.
6. Any history or evidence of tuberculosis (TB) (active or latent) using TB-QuantiFERON tests during screening.
7. Clinical signs and symptoms consistent with coronavirus disease 2019 (COVID-19).
8. Known history of primary immunodeficiency or an underlying condition that predisposes to infection.
9. Positive result for serum hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV).
10. Plasma donation within one month of the screening visit or any blood donation/blood loss > 500 mL during the 3 months prior to the screening visit.
11. Participants who have previously received AZD4144.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2025-04-23 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2025-06-27 (Actual)

PRIMARY OUTCOMES:
Area under concentration-time curve from time 0 to infinity (AUCinf) of AZD4144 | Days 1-4, Days 8-11 and Days 15-18
  1. To determine the relative bioavailability and compare the plasma exposure of AZD4144 in tablet formulation versus oral solution.
  2. To investigate the effect of a high-fat, high-calorie meal, in comparison to fasting conditions, on the PK of AZD4144 (dose 1 and dose 2) after a single oral tablet dose in healthy participants.
  3. To assess the effect of the proton pump inhibitor omeprazole on the PK of AZD4144 (dose 2) after a single dose.
Area under concentration-curve from time 0 to the last quantifiable concentration (AUClast) of AZD4144 | Days 1-4, Days 8-11 and Days 15-18
  1. To determine the relative bioavailability and compare the plasma exposure of AZD4144 in tablet formulation versus oral solution.
  2. To investigate the effect of a high-fat, high-calorie meal, in comparison to fasting conditions, on the PK of AZD4144 (dose 1 and dose 2) after a single oral tablet dose in healthy participants.
  3. To assess the effect of the proton pump inhibitor omeprazole on the PK of AZD4144 (dose 2) after a single dose.
Maximum observed drug concentration (Cmax) of AZD4144 | Days 1-4, Days 8-11 and Days 15-18
  1. To determine the relative bioavailability and compare the plasma exposure of AZD4144 in tablet formulation versus oral solution.
  2. To investigate the effect of a high-fat, high-calorie meal, in comparison to fasting conditions, on the PK of AZD4144 (dose 1 and dose 2) after a single oral tablet dose in healthy participants.
  3. To assess the effect of the proton pump inhibitor omeprazole on the PK of AZD4144 (dose 2) after a single dose.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | From Day 1 to Day 25
  To assess the safety and tolerability of single doses of AZD4144 in healthy participants.
Number of participants with serious AEs | From Screening (Day -28 to Day -2) to Day 25
  To assess the safety and tolerability of single doses of AZD4144 in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/